CLINICAL TRIAL: NCT05342324
Title: Optical Coherence Tomography Angiography in Choroidal Osteoma: a Quantitative Evaluation of Choriocapillary Vessel Density
Brief Title: Optical Coherence Tomography Angiography and Choroidal Osteoma
Status: Completed | Type: Observational
Sponsor: Federico II University (Other)
Responsible Party: Principal Investigator, Gilda Cennamo, Principal Investigator, Federico II University
Other Study IDs: 1604/21
Record Dates: First submitted 2022-04-16; First posted 2022-04-22 (Actual); Last update posted 2022-04-22 (Actual); Status verified 2022-04

CONDITIONS: Choroidal Osteoma, Bilateral
MeSH Terms: conditions — Choroidal Osteoma, Bilateral

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Optical coherence tomography angiography — To evaluate the vessel density in choriocapillary vascular networks, using optical coherence tomography angiography

SUMMARY:
This study evaluates the vessel density of choriocapillary vascular network in eyes affected by choroidal osteoma and in eyes complicated by choroidal neovascularization, using optical coherence tomography angiography.

DETAILED DESCRIPTION:
The choroidal osteoma is a rare benign tumor of choroid, it is bilateral in 10%-25% of cases, affecting usually young women. Previous studies evaluated the morphologic characteristics of tumor-related vasculatures, described as a seafun vascular networks, but none focused on study of vessel density of coriocapillary.

The aim of this study is to investigate the potential role of the optical coherence tomography angiography (OCTA) in evaluating the choriocapillary vessel density in order to individuate the changes of this vascular network that may influence the onset of choroidal neovasculariztion.

Therefore, OCTA could be useful in the clinical management of the choroidal osteoma

ELIGIBILITY:
Inclusion Criteria:

* age older than 50 years
* diagnosis of choroidal osteoma
* absence of history of vitreoretinal and vascular retinal diseases

Exclusion Criteria:

* age younger than 50 years
* no diagnosis of choroidal osteoma
* presence of history of vitreoretinal and vascular retinal diseases

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The participans were older than 50 years with choroidal osteoma. They did not present other ophthalmological diseases.
Sampling Method: Non-Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2015-06-01 (Actual); Primary Completion 2022-01-25 (Actual); Study Completion 2022-01-31 (Actual)

PRIMARY OUTCOMES:
Study of vessel density of the choriocapillary in patients affected by choroidal osteoma . | 7 years
  To evaluate the role of optical coherence tomography angiography in evaluating the features of the choriocapillary, using optical coherence tomography angiography (OCTA) in patients with choroidal osteoma and in patients with choroidal osteoma complicated by choroidal neovascularization. The parameter analyzed by OCTA was the vessel density of choriocapillary (percent)

CONTACTS AND LOCATIONS:
Overall Officials: Gilda Cennamo, Principal Investigator — Università Federico II
Locations (1):
- Federico II University, Naples, Napoli, Italy

REFERENCES:
- [Derived] Cennamo G, Iacucci G, Breve MA, Montorio D, Xompero C, Costagliola C. The role of choriocapillaris vessel density in the pathogenesis of macular neovascularization associated with choroidal osteoma. Graefes Arch Clin Exp Ophthalmol. 2023 May;261(5):1283-1287. doi: 10.1007/s00417-022-05921-1. Epub 2022 Dec 1. PMID 36454322